CLINICAL TRIAL: NCT02785458
Title: Testing a Medication Risk Communication and Surveillance Strategy: The EMC2 Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Boston Medical Center (Other); University of North Carolina, Chapel Hill (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Michael S. Wolf, Associate Division Chief - Research Division of General Internal Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00201638; 1R01DK103684 (NIH)
Record Dates: First submitted 2016-04-12; First posted 2016-05-27 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: High-risk Medications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Subjects will receive the current standard of care.
- EMC2 Strategy (Experimental): Subjects will receive the EMC2 Strategy. See description of strategy below.
  Interventions: Behavioral: EMC2 Strategy

INTERVENTIONS:
Behavioral: EMC2 Strategy — The intervention includes 1) distribution of simplified one-page medication guide summaries, 2) an automated follow-up call to assess medication safety and problematic side effects and 3) summary reports of call to providers with any concerns flagged for clinic follow-up.
  Arms: EMC2 Strategy

SUMMARY:
This study evaluates the effectiveness of an electronic health record based educational intervention (the EMC2 strategy) to improve patient understanding and use of higher-risk medications. Half of the participants will receive the intervention, while the other half will receive the usual amount of information (usual care).

DETAILED DESCRIPTION:
Research has repeatedly demonstrated that individuals lack essential information on how to safely take prescribed (Rx) medications. A risk communication and surveillance strategy is needed in primary care to ensure that patients are adequately informed about medication risks and are taking prescribed regimens safely.

The investigators devised an Electronic health record-based Medication Complete Communication (EMC2) Strategy that leverages electronic health record (EHR) and interactive voice response (IVR) technologies to:

1. prompt and guide provider counseling,
2. automate the delivery of Medication Guides at prescribing,
3. follow patients post-visit to confirm prescription understanding and use, and
4. deliver a care alert back to providers to inform them of any potential harms.

ELIGIBILITY:
Inclusion Criteria:

* 21 and older
* English or spanish speaking
* Primarily responsible for administering own medications
* New prescription of one of 66 study medications on day of recruitment
* Has a personal mobile or land line phone

Exclusion Criteria:

* Severe, uncorrectable vision
* Hearing or cognitive impairments

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Wolf, PhD, Principal Investigator — Northwestern University; Stacy C Bailey, PhD, Principal Investigator — Northwestern University; Michael K Paasche-Orlow, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Near North Health Services Corporation, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Usual Care | EMC2 Strategy
Started | 526 | 479
Completed | 526 | 479
Not Completed | 0 | 0
Period: 1 Month
Arm/Group | Usual Care | EMC2 Strategy
Started | 526 | 479
Completed | 443 | 404
Not Completed | 83 | 75
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 38 | 31
Not completed — Deemed Ineligible | 1 | 0
Not completed — Completed Evaluation by Baseline | 42 | 39
Not completed — Partial Interview | 0 | 4
Period: 3 Months
Arm/Group | Usual Care | EMC2 Strategy
Started | 443 | 404
Completed | 315 | 293
Not Completed | 128 | 111
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 25 | 21
Not completed — Completed Evaluation at 1 Month | 100 | 89

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | EMC2 Strategy | Total
Number analyzed (Participants) | 526 | 479 | 1005
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.34 (12.2) | 49.5 (12.6) | 50.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 319 | 299 | 618
  Male | 207 | 180 | 387
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 23 Individuals refused to identify their race, 4 individuals did not know how to identify their race
  Participants
    Race: number analyzed (Participants) | 515 | 463 | 978
    Race: Black or African American | 304 | 372 | 676
    Race: White | 78 | 35 | 113
    Race: Hispanic or Latino | 96 | 32 | 128
    Race: Others | 37 | 24 | 61
Education [Count of Participants; unit: Participants] — Population: 5 participants refused to answer the question, 1 did not know their highest education level
  Participants
    number analyzed (Participants) | 523 | 476 | 999
    Less than High School | 116 | 75 | 191
    High School Graduate | 292 | 318 | 610
    College Graduate | 115 | 83 | 198
Self-reported Health Status [Count of Participants; unit: Participants] — Population: 4 individuals refused to answer the question
  Participants
    number analyzed (Participants) | 524 | 477 | 1001
    Excellent/Very Good | 128 | 113 | 241
    Good | 179 | 177 | 356
    Fair/Poor | 217 | 187 | 404
Drug Class [Count of Participants; unit: Participants]
  Anticonvulsants | 123 | 95 | 218
  Antidepressants | 145 | 116 | 261
  Diabetes | 24 | 32 | 56
  LABA | 38 | 44 | 82
  NSAID | 59 | 61 | 120
  PPI | 25 | 27 | 52
  Others | 112 | 104 | 216
Preferred Language [Count of Participants; unit: Participants]
  English | 479 | 457 | 936
  Spanish | 47 | 22 | 69
Health Literacy (NVS) [Count of Participants; unit: Participants] — Health Literacy (NVS):Newest Vital Sign Population: 174 individuals did not complete the health literacy assessment
  Participants
    number analyzed (Participants) | 418 | 388 | 806
    Low | 172 | 177 | 349
    Marginal | 108 | 111 | 219
    Adequate | 138 | 100 | 238

OUTCOME MEASURES:

1. Primary Outcome: Medication Knowledge (0-100)
Description: Adjusted Least-square means of Medication Knowledge are calculated based on patient's ability to identify each medication's purpose and side effects, risks, warnings and benefits using general linear mixed models, specifying the identity link (PROC GLIMMIX). Treatment assignment by time is the independent variable of interest and modeled as a fixed effect, and clinic as a random effect, with additional subject statement to model correlations with patient. Confounding variables, such as age, preferred language, race, education, health status, number of chronic diseases, drug class, and health literacy (Newest Vital Sign) are included as fixed effects in the model. Patients are asked 10 questions (a scale developed by our team), and each questions is scored as correct/incorrect, and percentage of correctly answered questions is calculated (0-100 with 100 as best). Results are presented as adjusted least square means with 95% Confidence Intervals
Time Frame: Baseline to 3 Months post baseline
Population: 127 individuals were excluded from analysis, because their study med was either a short term medication or an antibiotics
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Usual Care | EMC2 Strategy
Number analyzed (Participants) | 459 | 419
score on a scale
  Baseline | 71.2 [68.5 to 73.9] | 71.9 [68.9 to 74.8]
  1 Month | 73.2 [70.5 to 75.9] | 74.9 [72.0 to 77.8]
  3 Months | 73.2 [70.4 to 75.9] | 75.0 [72.0 to 78.0]

2. Secondary Outcome: Probability of Prescription Medication Proper Use
Description: Subjects will be asked to demonstrate proper use of the medication by indicating the correct dose (amount of medication taken each time), frequency (times per day), and total pills/units per day. For non-PRN medications, all must be answered correctly to be considered proper use (yes/no) , whereas for PRN medications, proper use is determined if the patient indicated the correct dose or less, the correct frequency or less, and the correct total pills/units or less. Proper use is modelled as a binary outcome, and General linear mixed models are used, specifying the logit link (PROC GLIMMIX). Treatment assignment by time is the independent variable of interest and modeled as a fixed effect, and clinic as a random effect, with additional subject statement to model correlations with patient. Confounding factors, such as drug class and health literacy (Newest Vital Sign) are also included in the model as fixed effects. Results are presented as adjusted least square means with 95% CI
Time Frame: 1 Month post baseline to 3 Months post baseline
Population: 248 participants were excluded, due to either completing their evaluation early, or not filling their medication
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability
Arm/Group | Usual Care | EMC2 Strategy
Number analyzed (Participants) | 391 | 366
Probability
  1 Month | 0.84 [0.75 to 0.90] | 0.81 [0.71 to 0.88]
  3 Month | 0.83 [0.73 to 0.90] | 0.80 [0.68 to 0.88]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Usual Care | EMC2 Strategy
All-Cause Mortality (participants affected / at risk) | 0/526 | 0/479
Serious Adverse Events (participants affected / at risk) | 0/526 | 0/479
Other Adverse Events (participants affected / at risk) | 0/526 | 0/479

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT02785458/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT02785458/Prot_SAP_001.pdf